CLINICAL TRIAL: NCT00538096
Title: A Phase I, Multicenter, Open-Label, Single-Arm, Dose-Escalation, Study to Evaluate the Safety, Tolerability, and Antitumor Activity of Continuous Intravenous Infusion of the Bispecific T-Cell Engager MEDI-538 in Adults With B-Cell Non-Hodgkin's Lymphoma Not Eligible for Curative Therapy
Brief Title: A Phase I Study to Evaluate Safety, Tolerability in Adults With Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Replacing this trial with a new trial.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Karen L. Kaucic, M.D., MedImmune Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP137
Record Dates: First submitted 2007-09-28; First posted 2007-10-02 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Lymphoma, B-Cell; Lymphoma, Non-Hodgkin
Keywords: B-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): MEDI-538
  Interventions: Drug: MEDI-538
- 2 (Experimental): MEDI-538
  Interventions: Drug: MEDI-538
- 3 (Experimental): MEDI-538
  Interventions: Drug: MEDI-538

INTERVENTIONS:
Drug: MEDI-538 — 1 of 3 target doses of MEDI-538 (5,μg/m2/24h) as a continuous IV infusion through a central line catheter. The initial treatment period will be 4 weeks in duration (Study Days 0-27), unless the patient discontinues treatment.
  Arms: 1
Drug: MEDI-538 — 1 of 3 target doses of MEDI-538 (10,μg/m2/24h) as a continuous IV infusion through a central line catheter. The initial treatment period will be 4 weeks in duration (Study Days 0-27), unless the patient discontinues treatment.
  Arms: 2
Drug: MEDI-538 — 1 of 3 target doses of MEDI-538 (15,μg/m2/24h) as a continuous IV infusion through a central line catheter. The initial treatment period will be 4 weeks in duration (Study Days 0-27), unless the patient discontinues treatment.
  Arms: 3

SUMMARY:
* Evaluate the safety and tolerability of multiple doses of MEDI-538 by continuous IV infusion for 4 or 8 weeks in adult patients with B-cell NHL not eligible for curative therapy.
* Determine the maximum tolerated dose of MEDI-538 administered by continuous IV infusion.

DETAILED DESCRIPTION:
* Evaluate the safety and tolerability of MEDI-538 at doses of 5, 10, or 15 μg/m2/24h by continuous IV infusion for 4 or 8 weeks in adult patients with B-cell NHL not eligible for
* Determine the MTD of MEDI-538 administered by continuous IV infusion for 4 or 8 weeks in adult patients with B-cell NHL not eligible for curative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women at least 18 years of age;
* Written informed consent and Heath Insurance Portability and Accountability Act (HIPAA) authorization (applies to covered entities in the US only) obtained from the patient prior to performing any study-related procedures, including screening visits;
* Histologically confirmed B-cell NHL of one of the following classifications:

  * Follicular lymphoma
  * Marginal zone lymphoma;
  * Lymphoplasmocytic lymphoma; or
  * Mantle cell lymphoma.
* Not eligible for curative therapy according to the NCCN guidelines for NHL (NCCN 2006);
* Measurable disease (at least one lesion ≥ 20 mm in one dimension) documented by computed tomography (CT) scan;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (see Appendix A);
* Life expectancy of at least 6 months;
* Heterosexual sexually active females, unless surgically sterile or at least 1 year postmenopausal, must use an effective method of avoiding pregnancy (including oral or implanted contraceptives, intrauterine device, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) for 21 days prior to the first dose of study drug, and must agree to continue using such precautions through 3 months after the last dose of MEDI-538. Cessation of birth control after this point should be discussed with a responsible physician. Heterosexual sexually active males, unless surgically sterile, must likewise use an effective method of birth control (condom) and must agree to continue using such precautions through 3 months after the last dose of MEDI-538;
* Hemoglobin ≥ 10.0 g/dL; absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L; platelets ≥ 100.0 × 10^9/L; lymphocyte count ≥ 0.8 × 10^9/L; leukocyte count ≥ 3.0 × 10^9/L; and D-dimer ≤ 2.5 × upper limit of normal (ULN); and antithrombin III ≥ lower limit of normal (LLN); and 10. Total bilirubin ≤ 1.5 × ULN; aspartate transaminase (AST), alanine transaminase (ALT), amylase and lipase ≤ 2 × ULN; serum creatinine ≤ 2 × ULN, and creatinine clearance ≥ 50 mL/min.

Exclusion Criteria:

* Receipt of MEDI-538 in any previous clinical study;
* History of allergy or reaction to any component of the MEDI-538 formulation;
* Any other NHL not listed in inclusion criterion 3;
* History of malignancy other than B-cell NHL within 5 years prior to study entry, with the exception of basal cell carcinoma of the skin or carcinoma in situ of the cervix successfully treated with curative therapy;
* Known or suspected CNS involvement by NHL;
* Clinical history of significant CNS pathology, eg, multiple occurrences of confusion, dementia, multiple previous infarcts, or major brain surgery;
* Active infection or known bacteremia. Patients with documented evidence of culture positive sepsis or active infection requiring IV antibiotic therapy must complete a full course of antibiotic treatment with no clinical or laboratory evidence of bacterial infection at least 2 weeks prior to starting therapy with MEDI-538.
* Vaccination (either preventive or therapeutic for infectious disease or cancer) within 2 weeks prior to initiation of study drug;
* Infection with human immunodeficiency virus (HIV-1 or HIV-2), chronic infection with hepatitis B or C, or acute infection with hepatitis A;
* History of primary immunodeficiency;
* History of serious, chronic autoimmune disease, eg, rheumatoid arthritis, systemic lupus erythematosus, and multiple sclerosis;
* Elective surgery planned during the study period through 30 days after discontinuation of MEDI-538;
* Autologous stem cell transplantation within 26 weeks prior to study entry;
* Allogenic stem cell transplantation or any other solid organ transplant;
* Cancer chemotherapy within 6 weeks prior to study entry;
* Radiotherapy within 6 weeks prior to study entry;
* Receipt of any investigational agent within 12 weeks prior to initiation of study drug;
* Treatment with rituximab within 12 weeks prior to study entry;
* Prior treatment with alemtuzumab;
* Regular dose of systemic corticosteroids during the 4 weeks prior to initiation of study drug or anticipated need of corticosteroids exceeding prednisone 20 mg/day or equivalent during the trial, or any other systemic immunosuppressive therapy within 4 weeks prior to study entry;
* Any contraindication to chronic anticoagulation with low-molecular weight heparin (LMWH);
* Inability for safe placement and prolonged use (at least 8 weeks) of a central venous catheter;
* Contraindication to any of the protocol-specified concomitant medications (methylprednisolone, antacids, or antihistamines) during this study;
* Presence of human anti-murine antibodies or known hypersensitivity to immunoglobulins;
* Pregnancy (sexually active females of childbearing potential must have a negative urine pregnancy test on the day of the first dose of the study drug, prior to dosing) or nursing;
* Evidence of any uncontrolled systemic disease (other than B-cell NHL), any finding upon physical examination or history of any disease that, in the opinion of the investigator or medical monitor, may compromise the safety of the patient in the study or confound the analysis of the study; or
* Inability to meet social environment requirements for outpatient therapy (see Section 3.3.4.4).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-03 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
All endpoints will be analyzed descriptively. AEs and SAEs will be summarized by dose cohort, body system, severity, and relationship to MEDI-538 through 30 days after discontinuation of MEDI-538. | 30 days after discontinuation of MEDI-538

SECONDARY OUTCOMES:
The secondary endpoints of this study include measurement of the pharmacokinetics,immunogenicity, and antitumor activity of MEDI-538 in this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Karen L. Kaucic, M.D., Study Director — MedImmune LLC